CLINICAL TRIAL: NCT05983588
Title: Double-blind, Randomised, Prospective, Placebo Controlled Parallel Group Phase II Study to Investigate the Effect of Glycerol Phenylbutyrate (GPB) on Neurofilament Light Chain (NfL) Levels in Patients With Corticobasal Syndrome (CBS)
Brief Title: PROFIL Study to Investigate the Effect of GPB on NfL Levels in Patients With Corticobasal Syndrome (CBS)
Acronym: PROFIL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PROFIL-2088-SIM-0032-I
Record Dates: First submitted 2023-07-13; First posted 2023-08-09 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-08

CONDITIONS: Corticobasal Syndrome (CBS)
MeSH Terms: conditions — Corticobasal Degeneration | interventions — glycerol phenylbutyrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verum (Experimental): RAVICTI 1.1 g/ml oral liquid (glycerol phenylbutyrate (GPB)) Duration of Treatment: 26 weeks, twice daily
  Interventions: Drug: RAVICTI 1.1 g/ml
- Placebo (Placebo Comparator): Matching Placebo, oral liquid Duration of Treatment: 26 weeks, twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RAVICTI 1.1 g/ml — Duration of Treatment: 26 weeks, twice daily
  Dosage:
  * weeks 0 - 3: 3 ml/day (1,5ml - 0 - 1,5ml) (≙ 3,3 g glycerol phenylbutyrate/placebo)
  * weeks 4 - 26: 6 ml/day (3 ml - 0 - 3 ml) (≙ 6,6 g glycerol phenylbutyrate/placebo)
  Other Names: Glycerol phenylbutyrate
  Arms: Verum
Drug: Placebo — Duration of Treatment: 26 weeks, twice daily
  Dosage:
  * weeks 0 - 3: 3 ml/day (1,5ml - 0 - 1,5ml) (≙ 3,3 g glycerol phenylbutyrate/placebo)
  * weeks 4 - 26: 6 ml/day (3 ml - 0 - 3 ml) (≙ 6,6 g glycerol phenylbutyrate/placebo)
  Arms: Placebo

SUMMARY:
Corticobasal syndrome (CBS) is a rapidly progressive neurodegenerative disorder with an average survival time of about 6-8 years after the first clinical manifestation. No potent symptomatic treatment is currently available. A disease-modifying therapy does not exist either. Neuroinflammation is key to the pathogenesis in neurodegenerative diseases with Tau- and/or AD-pathology. There is strong evidence that phenylbutyrate can modulate microglial function by enhancing their phagocytic activity, most likely by epigenetic mechanisms. So the main goal of this clinical trial is to study a potential disease-modifying effect of treatment with glycerol phenylbutyrate (GPB), which is a prodrug of phenylbutyric acid, for 26 weeks assessed by the levels of the biomarker neurofilament light chain (NfL) indicating disease progression in CBS. Given the aggressive nature of CBS, it is feasible to study effects of GPB on plasma NfL levels.

ELIGIBILITY:
Inclusion Criteria:

1. Age: ≥ 18 years
2. "clinical possible" or "clinical probable" CBS (Armstrong et al., Neurol-ogy, 2013 80;496-503) and patients with Progressive Supranuclear Palsy-CBS according to Höglinger et al. (Mov Disord. 2017 Jun;32(6):853-864)
3. No regular consumption of glycerol phenylbutyrate within the last 6 months prior to V1
4. Capable of thoroughly understanding all information given and giving full informed consent according to GCP
5. Capability and willingness to comply with the procedures of the clinical trial
6. Women of childbearing age must be non-lactating and surgically sterile or using a highly effective method of birth control and have a nega-tive pregnancy test. In case of using a hormonal contraception, the method must be supplemented with a barrier method (preferably male condom). Acceptable methods of birth control with a low failure rate i.e. less than 1% per year when used consistently and correct are such as implants, injectables, combined oral contraceptives, hormonal intrauterine devices (IUDs), sexual abstinence (defined as refraining from heterosexual intercourse during the clinical trial) or vasectomized partner. Unacceptable birth control methods are: periodic abstinence (calendar, symptothermal, post-ovulation methods), withdrawal (coitus interruptus), spermicides only and lactational amenorrhoea method (LAM). Female condom and male condom should not be used together.
7. A stable regimen for at least 1 month prior to V1 and no foreseeable need to change the regimen throughout the 26 week treatment period for

   1. drugs acting against Parkinsonism (e.g. Levodopa, Dopamine-Agonists, Amantadine and MAO-B-Inhibitors)
   2. other CNS-active substances including e.g. antidepressants and antidementia drugs

Exclusion Criteria:

1. Neurodegenerative diseases other than CBS
2. Underlying Alzheimer's pathology as defined by positive β-amyloid-PET or reduced Aβ 1-42 in CSF
3. Participation in another clinical trial involving administration of an investigational medicinal product within 1 month or 5 half-lives of the investigational medicinal product, whichever is longer, prior to V1
4. Known hypersensitivity to glycerol phenylbutyrate or its further components, or to drugs with a similar chemical structure or to any of the components of the placebo
5. Treatment with valproic acid, haloperidol or probenecid
6. A physical or psychiatric condition (e.g. frontal lobe syndrome, psychotic disorder or major depression), which at the investigator's discretion may put the subject at risk, may confound the trial results or may interfere with the subject's participation in this clinical trial
7. Persistent abuse of medication, drugs or alcohol
8. Current or planned pregnancy or breast-feeding in females
9. Other severe medical conditions upon the discretion of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
To assess the efficacy of glycerol phenylbutyrate vs. placebo in reducing the levels of neurofilament light chain (NfL) during 26 weeks of exposure to glycerol phenylbutyrate as well as safety and tolerability of glycerol phenylbutyrate in patients with | 26 weeks (between V1 and V3)
  To assess the efficacy of glycerol phenylbutyrate vs. placebo in reducing the levels of neurofilament light chain (NfL) during 26 weeks of exposure to glyc-erol phenylbutyrate as well as safety and tolerability of glycerol phenylbutyrate in patients with CBS.

SECONDARY OUTCOMES:
To assess longitudinal changes in clinical scales | 26 weeks (between V1 and V3)
  To assess longitudinal changes in clinical scale: Movement Disorder Society Unified Parkinson's Disease Rating Scale (MDS-UPDRS Part III), min value 0- max value 132 (worse outcome)
To assess longitudinal changes in clinical scales | 26 weeks (between V1 and V3)
  To assess longitudinal changes in clinical scale: Progressive Supranuclear Palsy Rating Scale (PSP-RS), min value 0- max value 100 (worse outcome)
To assess longitudinal changes in clinical scales | 26 weeks (between V1 and V3)
  To assess longitudinal changes in clinical scale:Progressive Supranuclear Palsy Clinical Deficits Scale (PSP-CDS), min value 0- max value 21 (worse outcome)
To assess longitudinal changes in clinical scales | 26 weeks (between V1 and V3)
  To assess longitudinal changes in clinical scale: Cortical Basal ganglia Functional Scale (CBFS), min value 0- max value 124 (worse outcome)
To assess longitudinal changes in clinical scales | 26 weeks (between V1 and V3)
  To assess longitudinal changes in clinical scale: Dementia Apraxia Test (DATE), min value 0 (worse outcome) - max value 60
To assess longitudinal changes in clinical scales | 26 weeks (between V1 and V3)
  To assess longitudinal changes in clinical scale: MONTREAL COGNITIVE ASSESSMENT (MoCA), min value 0 (worse outcome) - max value 30
To assess longitudinal changes in clinical scales | 26 weeks (between V1 and V3)
  To assess longitudinal changes in clinical scale: SCHWAB AND ENGLAND ACTIVITIES OF DAILY LIVING SCALE (SEADL), min value 0 (worse outcome) - max value 100%
To assess longitudinal changes in clinical scales | 26 weeks (between V1 and V3)
  To assess longitudinal changes in clinical scale: Clinical Global Impression (CGI-s), min value 1- max value 7 (worse outcome)
To assess longitudinal changes in clinical scales | 26 weeks (between V1 and V3)
  To assess longitudinal changes in clinical scale: PSP RATING SCALE (PSP-QoL), min value 0- max value 180 (worse outcome)

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Klinikum der Universität München (KUM), Campus Großhadern, Klinik und Poliklinik für Neurologie & German Center for Neurodegenerative Diseases (DZNE), Department of Neurology, Munich, Bavaria
  - Klinikum rechts der Isar Technische Universität München Klinik und Poliklinik für Neurologie & German Center for Neurodegenerative Diseases (DZNE), Department of Neurology, Munich, Bavaria

IPD SHARING:
Plan to Share IPD: No